CLINICAL TRIAL: NCT02404116
Title: Metacognitive Therapy for Health Anxiety: A Randomised Control Trial
Brief Title: Metacognitive Therapy for Health Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Robin Bailey, Principal Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: : z83hdhmg
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Hypochondriasis
MeSH Terms: conditions — Hypochondriasis | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metacognitive Therapy (Experimental): 12 weeks of Metacognitive Therapy
  Interventions: Other: Metacognitive Therapy
- Wait List Control (Other): The Waiting list control will control for time and repeated assessments during an initial 12 week period
  Interventions: Other: Wait List

INTERVENTIONS:
Other: Metacognitive Therapy — Participants will receive treatment which focus's on helping reduce excessive thinking about health,
  Arms: Metacognitive Therapy
Other: Wait List — Individuals are on a waiting list
  Arms: Wait List Control

SUMMARY:
The study involves a comparing a new psychological treatment- Metacognitive Therapy (MCT) which has shown promising results in the treatment of health anxiety to no treatment at all- a waiting list.

DETAILED DESCRIPTION:
Hypochondriasis or severe health anxiety is characterised by excessive, disproportionate and persistent thoughts, behaviour and emotion focused on physical symptoms and/or fear of developing a serious illness. There is often excessive worry about illness or disease in the absence of supporting medical evidence and contrary to continual medical reassurance.

The most effective psychological treatments are cognitive and behavioural therapies (CBT). However, CBT has failed to demonstrate consistent gains in the treatment of this disorder.

A newer form of psychological therapy, Metacognitive Therapy (MCT) has shown to be more effective than CBT in the treatment of anxiety disorders and depression. MCT is based on the principle that health anxiety is caused by a pattern of extended thinking, this pattern is called the Cognitive Attentional Syndrome (CAS). The CAS is made up of chains of verbal thought in the form of excessive worry about having an illness; a pattern of focusing attention on threat, such as scanning the body for signs of illness and excessive body checking; and coping strategies that have negative effects, such as internet searching for illnesses or trying to block out thoughts of illness. Rather than stopping negative thinking the CAS extends it and leads to the belief that illness is present. To help reduce these symptoms MCT teaches specific techniques that help people develop new ways of experiencing negative thoughts about illnesses, allow them to abandon worry and learn to disengage from unhelpful coping attempts.

A recent small study has provided some limited evidence that metacognitive therapy (MCT) can be applied to cases of hypochondriasis and demonstrated that the therapy was associated with improvement in symptoms.

To provide future evaluation of MCT in this client group a more definitive trial will be carried out to ascertain the effects of MCT in a larger group when compared to a control group.

If the results are positive this will provide a rationale for a larger research study, which will compare MCT with evidence based treatment such as CBT.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18.
* Exceed cut off on BP and WI
* Not undergoing any other form of psychological therapy during treatment.
* If on medication must be stable six weeks prior to treatment onset.
* Willing to undergo randomisation
* Provide written consent

Exclusion Criteria:

* Be under 18
* Not exceeding cut off on BP and WI
* Undergone CBT for health anxiety over the past three months.
* Having started medication less than four weeks before assessment
* Not willing to undergo randomisation
* Not willing to provide written consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in health anxiety levels over 12weeks of treatment measured by the Whiteley Index 7 (WI7) | This will be administered in the first and last treatment session (week 1 and week 12) by the study investigators, and once at 6 months follow up following treatment completion
  Measures the presence of health anxiety.
Change in health anxiety levels over 12weeks of treatment measured by the Bodily Perception Questionnaire (BP). | This will be administered in the first and last treatment session (week 1 and week 12) by the study investigators, and once at 6 months follow up following treatment completion
  Measures the presence of health anxiety.

SECONDARY OUTCOMES:
Change in anxiety levels over 12weeks of treatment measured by the Beck Anxiety Inventory | This will be administered in the first and last treatment session (week 1 and week 12) by the study investigators, and once at 6 months follow up following treatment completion
  Will be used as a measure of anxiety
Change in general metacognition levels over 12weeks of treatment measured by the The Metacognitions Questionaire-30 (MCQ-30) | This will be administered in the first and last treatment session (week 1 and week 12) by the study investigators, and once at 6 months follow up following treatment completion
  will be used to examine general positive and negative beliefs about worrying thoughts, attitudes & processes.
Change in depression levels over 12weeks of treatment measured by the Beck Depression inventory | This will be administered in the first and last treatment session (week 1 and week 12) by the study investigators, and once at 6 months follow up following treatment completion
  Will be used as general mood measures
Change in health anxious metacognition levels over 12weeks of treatment measured by the The Meta-Cognitions about Health Questionnaire (MCHQ) | This will be administered in the first and last treatment session (week 1 and week 12) by the study investigators, and once at 6 months follow up following treatment completion
  Specific metacognitive beliefs associated with health anxiety
Change in dysfunctional beliefs over 12weeks of treatment measured by the Health cognition Questionnaire | This will be administered in the first and last treatment session (week 1 and week 12) by the study investigators, and once at 6 months follow up following treatment completion
  Dysfunctional beliefs associated with health anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Robin Bailey, MSc, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - University of Central Lancashire, Preston, Lancashire
  - University of Manchester, Manchester, Manchester